CLINICAL TRIAL: NCT02207595
Title: A Randomized, Investigator- and Subject-blind, Placebo-controlled, Combined Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles of UCB5857 in Healthy Subjects
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles of UCB5857 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Celltech (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP0021; 2014-002361-30 (EudraCT Number)
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- UCB5857 Cohort 1 (Experimental): UCB5857 and Placebo: Single dose followed by multiple doses over 14 days
  Interventions: Drug: UCB5857; Other: Placebo
- UCB5857 Cohort 2 (Experimental): UCB5857 and Placebo: Single dose followed by multiple doses over 14 days
  Interventions: Drug: UCB5857; Other: Placebo
- UCB5857 Cohort 3 (Experimental): UCB5857 and Placebo: Single dose followed by multiple doses over 14 days
  Interventions: Drug: UCB5857; Other: Placebo
- UCB5857 Cohort 4 (Experimental): UCB5857 and Placebo: Single dose followed by multiple doses over 14 days
  Interventions: Drug: UCB5857; Other: Placebo
- UCB5857 Cohort 5 (Experimental): UCB5857 and Placebo: Single dose followed by multiple doses over 14 days
  Interventions: Drug: UCB5857; Other: Placebo

INTERVENTIONS:
Drug: UCB5857 — * Active Substance: UCB5857
  * Pharmaceutical Form: Capsule
  * Concentrations: 5 mg, 10 mg, 20 mg, 30 mg, 50 mg, 100 mg
  * Route of Administration: Oral Use
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Capsule
  * Concentrations: 5 mg, 10 mg, 20 mg, 30 mg, 50 mg, 100 mg
  * Route of Administration: Oral Use

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of UCB5857.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, all of the following criteria must be met:

* An Independent Ethics Committee (IEC)-approved written Informed Consent Form is signed and dated by the subject
* Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, or medication intake according to the judgment of the Investigator
* Subject is male or female, 18 to 55 years of age (inclusive)
* Female subjects must have a negative pregnancy test in urine at the Screening Visit and a negative serum pregnancy test on Day -1, and be of nonchildbearing potential, defined as being:

  1. Postmenopausal (for at least 2 years before the Screening Visit), verified by serum follicle-stimulating hormone (FSH) level >40 mIU/mL at the Screening Visit, or
  2. Permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy), or
  3. Congenitally sterile
* Contraception methods for male subjects and their female partners:

  1. Male subject with a partner of childbearing potential must be willing to use a condom when sexually active
  2. The female partner of childbearing potential of a male subject must be willing to use at least 2 effective methods of contraception, including a barrier method (eg, male condom, female condom, or diaphragm with spermicide) during the study period.

Both sexes must use the above mentioned contraception methods (condoms for males) during the study and for 20 weeks after the last administration of the Investigational Medicinal Product (IMP) (anticipated 5 half-lives).

* Subject is of normal weight as determined by a body mass index (BMI) of 18.0 to 30.0 kg/m^2 (inclusive), with a body weight of at least 50 kg
* Subject has clinical laboratory test results within the reference ranges of the testing laboratory
* Subject has Blood Pressure (BP) and pulse within normal range in a supine position after 5 minutes rest (systolic BP: 90 to 140 mmHg, diastolic BP: 50 to 90 mmHg, pulse: 40 to 90 beats per minute - all inclusive)
* Subject's ECG is considered "normal" or "abnormal but clinically nonsignificant" (as interpreted by the Investigator)

Exclusion Criteria:

Subjects are not permitted to enroll in the study if any of the following criteria is met:

* Subject has a known hypersensitivity to any components of the Investigational Medicinal Product (IMP)
* Subject is considered anti-high-affinity immunoglobulin E (IgE) receptor nonresponsive if CD63 induction on basophils is <10 %
* Subject has cardiovascular or cerebrovascular disease, including hypertension, angina, ischemic heart disease, transient ischemic attacks, stroke, and peripheral arterial disease sufficient to cause symptoms and/or require therapy to maintain stable status
* Subject has diabetes mellitus of any type requiring insulin
* Subject has

  1. an active infection (eg, sepsis, pneumonia, abscess)
  2. history of latent, chronic, or recurrent infections (eg, tuberculosis [TB], recurrent sinusitis, genital herpes, urinary tract infections) or at risk of infection (surgery, trauma, infection requiring antibiotics, history of skin abscesses) within 3 months before IMP administration
  3. experienced a significant episode of gastroenteritis (defined as loose stools associated with abdominal pain and/or fever) during the 7 days before IMP administration

When in doubt, the Investigator should confer with the Sponsor's Study Physician.

* Subject has a history of positive TB test or evidence of possible TB or latent TB infection at the Screening Visit (QuantiFERON® Gold Test)
* Subject has received live attenuated vaccination within 3 months or any other type of vaccine within 4 weeks before the Screening Visit or intends to have such a vaccination during the course of the study
* Subject who has any of the following hematology values at the Screening Visit: Hemoglobin; for women <11 g/dL; for men <13 g/dL Absolute Neutrophil Count (ANC) <1.5 x 109/L (<1000/mm^3)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events during the study | Day -1 to multiple dose Day 17

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC(0-24)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
Area under the plasma concentration-time curve from time 0 to infinity (AUC) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
The maximum observed plasma concentration of UCB5857 after single dosing, obtained directly from the observed plasma concentration-time curves (Cmax) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
The time of occurrence of Cmax, obtained directly from the observed plasma concentration-time curves (tmax) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
The apparent terminal half-life (t1/2) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
The terminal elimination rate constant in plasma (λz) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
The apparent volume of distribution after single dosing (Vz/F) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
The apparent total body clearance after single dosing (CL/F) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
Mean residence time (MRT) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC(0-24)) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The time of occurrence of Cmax, obtained directly from the observed plasma concentration-time curves (tmax) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The apparent terminal half-life (t1/2) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The terminal elimination rate constant in plasma (λz) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
Mean residence time (MRT) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The apparent volume of distribution at steady state (Vzss/F) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The apparent total body clearance at steady state (CLss/F) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The maximum observed plasma concentration of UCB5857 during steady state, obtained directly from the observed plasma concentration-time curves (Cmaxss) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
The minimum observed plasma concentration of UCB5857 during steady state immediately before the next dose would be administered, obtained directly from the observed plasma concentration-time curves (Ctrough) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
Accumulation factor based on AUC(0-24) (RAUC) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
Accumulation factor based on Cmax (R(Cmax)) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
Time independency factor (TI) | Pharmacokinetic samples will be taken predose on MD-Days 1 to 13, predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours postdose on MD-Day 14, 24 hours postdose (MD-Day 15), 48 hours postdose (MD-Day 16) and 72 hours postdose (MD-Day 17)
Basophil degranulation | Samples will be taken at Screening, SD-Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10 hours postdose) and 24, 48 hours postdose. Samples will also be taken on MD-Days 4, 8 , 13 at predose, 0.25, 0.5, 1, 2, 4, 6, 8 and 10 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Harrow, United Kingdom